CLINICAL TRIAL: NCT01958866
Title: Study of Efficacy and Safety of Tinospora Crispa-extract Product Compared With the Acetaminophen
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Pornanong Aramwit, Pharm.D., Ph.D, Associate Professor, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0156
Record Dates: First submitted 2013-09-11; First posted 2013-10-09 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-03

CONDITIONS: Patients With Body Temperature Between 37.8-38.5; No Sign of Infection; No Liver and Kidney Problem
Keywords: Fever; Body temperature
MeSH Terms: conditions — Fever | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Acetaminophen (Active Comparator): Acetaminophen administer 1000 mg every 4-6 hours when fever is presented
  Interventions: Drug: Acetaminophen
- Tinospora Crispa-extract Product (Experimental): Tinospora Crispa-extract tablet administer 500 mg every 4-6 hours when fever is presented
  Interventions: Drug: Tinospora Crispa-extract Product
- Placebo (Placebo Comparator): Placebo 2 tablets will be administered every 4 hours when fever is presented
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Tinospora Crispa-extract Product
  Arms: Tinospora Crispa-extract Product
Drug: Acetaminophen
  Arms: Acetaminophen
Other: Placebo
  Arms: Placebo

SUMMARY:
Hypothesis: Tinospora Crispa-extract Product can reduce pyretic similar to acetaminophen.

This study aims to investigate the efficacy and safety of Tinospora Crispa-extract product compared with the acetaminophen. Total of 96 patients with body temperature between 37.8-38.5 without any signs of infections will be enrolled in this study. Patients will be randomly divided into 3 groups: First group will receive acetaminophen 1000 mg every 6 hr, Second group will receive Tinospora Crispa-extract Product 2000 mg twice daily and the third group will receive placebo twice daily.

DETAILED DESCRIPTION:
Patients in each group will be monitored for body temperature at baseline (at the time of enrollment) and at 1, 2, 4, 6, 8, 24 h after receiving the tested material.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years old
* Body temperature between 37.8-38.5
* Body weight not less than 40 kg but not over 100 kg
* Liver enzymes do not exceed 2 times of normal value
* Can comply with study protocol

Exclusion Criteria:

* Have allergic history of any tested compounds
* Fever from other causes, not by URI
* Take any herbal medicines during 2 weeks before enrollment
* Physicians decide to withdraw the subjects with any reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2013-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Body Temperature | Change from baseline in temperature at 1, 2, 3, 4, 6, 8, 12 and 24 hours

SECONDARY OUTCOMES:
Number of adverse events: diarrhea, elevated liver enzyme and elevated creatinine | Participants will be followed for the duration of hospital stay (24 hours)
  Liver and kidney function will be randomly evaluated. Number of participants with soft stool will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Pornanong Aramwit, Bangkok, Bangkok, Thailand